CLINICAL TRIAL: NCT03880149
Title: The Effects of Omega-3 Status and Supplementation on Tendon Structure and Recovery From Sports Injuries in Competitive Athletes
Brief Title: The Effects of Omega-3 Status and Supplementation on Tendon Structure in Competitive Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: University of Haifa (Other); Tel Hai College (Other)
Responsible Party: Principal Investigator, Dan Nemet, MD, Professor of Pediatrics. Director, Child Health and Sports Center, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MeirMc0242-18CTIL
Record Dates: First submitted 2018-12-02; First posted 2019-03-19 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Tendon Injuries; Inflammation
Keywords: Omega-3; Athletes; Sports injuries; Inflammatory markers; Isokinetic muscle force
MeSH Terms: conditions — Tendon Injuries; Inflammation; Athletic Injuries | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 supplementation (Experimental): Omega-3 fatty supplementation and vitamin E. Each 1 g omega-3 capsule contain 600 mg omega-3 including 400 mg EPA + 200 mg DHA. Individual omega-3 dose will be determined according to the athlete's body mass, 1 g omega-3 / 15 kg body mass per day and vitamin E: 1 capsule of vitamin E (400 IU) for every five omega-3 capsules
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): Medium-chain triglyceride (MCT) and vitamin E. Each MCT capsule contain 1 g, the dose will be 115 mg per kg body mass per day, and vitamin E: 1 capsule of vitamin E (400 IU) for every five MCT capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — Each omega-3 capsule contains 600 mg, including 400 mg EPA + 200 mg Docosahexaenoic acid (DHA) and 400 IU of vitamin E for 5 omega-3 capsules. Omega-3 dosage: 1 g per 15 kg body mass
  Arms: Omega-3 supplementation
Other: Placebo — Medium-chain triglyceride (MCT) and vitamin E
  Arms: Placebo

SUMMARY:
The study will examine the association between omega-3 status and the effects of omega-3 supplementation on changes in tendon structure and recovery from tendon injuries and inflammatory markers in competitive athletes. Half of the participants will receive omega-3 in combination with vitamin E, while the other half will receive a placebo and vitamin E.

DETAILED DESCRIPTION:
Sports injuries are common among athletes, while injury prevention received much clinical attention, there is no consensus among clinicians and researchers as to which injury-causing factors are dominant. It has been suggested that increased training load may be the leading cause of sports injuries, since tendons are sensitive to changes in load, making them vulnerable to injury. Inflammation is one of the reversible risk factors to sports injuries, and there are numerous methods which are used to treat inflammation. It has been recently suggested that inflammation reactions are affected by Omega-3 status and that omega-3 deficiency may increase the risk of sports and tendon injuries. The omega-3 fatty acid may act as a regulator of membrane structure and function, intracellular signaling pathways, transcription factor activity, and gene expression and reducing inflammation. Due to these functions, omega-3 may influence exercise-induced injuries/inflammation in athletes, thus, may influence their health and allowing training.

ELIGIBILITY:
Inclusion Criteria:

Part one:

* Training for at least 5 hours per week.
* No complaints about lower extremities pains during the last 12 months.

Part two:

* Training for at least 5 hours per week.
* Diagnosed with patellar and Achilles tendinitis.

Exclusion Criteria:

* Underwent lower extremities surgeries.
* Allergic to Fish products.
* Athletes who use anti-inflammatory drugs and/or omega-3 supplements.
* Pregnant and/or nursing mothers.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Tendon Structure | 6 months
  Changes in the echo pattern of patellar and Achilles tendons structure using Ultrasound Tissue Characterization (UTC). Distribution (%) of echo type 1-3.

SECONDARY OUTCOMES:
Inflammatory marker | 3 months
  Serum interleukin 6 (IL-6) (pg/mL)
Muscle Strength | 6 months
  Total work (Kjoule) (using Biodex isokinetic testing protocol)
Omega-3 status | 6 months
  Distribution (%) of 26 identified fatty acids - measured in Blood
Cross sectional area of Achilles tendon | 6 months
  measured using Ultrasound Tissue Characterization (UTC) (cm^2)
Range of motion - knee | 6 months
  using digital inclinometer for range of motion measurement (degrees)
Pain assessment | 6 months
  pain severity using visual analog scale (VAS) - on a scale of 0 -10, 0 being no pain and 10 the worst pain ever
functional assessment | 3 months
  VISA P questionnaire - scale 0-100
Pro-inflammatory cytokine. | 3 months
  Serum interleukin 17 (IL-17) (pg/mL)
Marker for inflammation | 3 months
  C Reactive Protein (CRP) (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center, Kfar-Saba, Israel; Gali Dar, PhD, Study Director — University of Haifa; Yitzhak Weinstein, PhD, Study Director — Tel Hai Academic College
Locations (1):
- Wingate institute, Netanya, Israel

REFERENCES:
- [Background] Da Boit M, Hunter AM, Gray SR. Fit with good fat? The role of n-3 polyunsaturated fatty acids on exercise performance. Metabolism. 2017 Jan;66:45-54. doi: 10.1016/j.metabol.2016.10.007. Epub 2016 Oct 26. PMID 27923448
- [Result] Black KE, Witard OC, Baker D, Healey P, Lewis V, Tavares F, Christensen S, Pease T, Smith B. Adding omega-3 fatty acids to a protein-based supplement during pre-season training results in reduced muscle soreness and the better maintenance of explosive power in professional Rugby Union players. Eur J Sport Sci. 2018 Nov;18(10):1357-1367. doi: 10.1080/17461391.2018.1491626. Epub 2018 Jul 9. PMID 29985775
- [Result] Lewis EJ, Radonic PW, Wolever TM, Wells GD. 21 days of mammalian omega-3 fatty acid supplementation improves aspects of neuromuscular function and performance in male athletes compared to olive oil placebo. J Int Soc Sports Nutr. 2015 Jun 18;12:28. doi: 10.1186/s12970-015-0089-4. eCollection 2015. PMID 26085822
- [Result] von Schacky C, Kemper M, Haslbauer R, Halle M. Low Omega-3 Index in 106 German elite winter endurance athletes: a pilot study. Int J Sport Nutr Exerc Metab. 2014 Oct;24(5):559-64. doi: 10.1123/ijsnem.2014-0041. Epub 2014 Sep 8. PMID 25203220